CLINICAL TRIAL: NCT01159470
Title: CRP Velocity as a Marker for Bacterial Infections in Children
Brief Title: The Rate of C-reactive Protein (CRP) Increase as a Marker for Bacterial Infections in Children
Acronym: CRPv
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Maskit Bar-Meir, MD, Shaare-Zedek Medical Center
Other Study IDs: 472010.ctil
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Bacterial Infections; Viral Infection
Keywords: CRP velocity
MeSH Terms: conditions — Bacterial Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- bacterial infection: children with fever due to bacterial infection
- viral infection: children with fever due to viral infection

SUMMARY:
Fever is one of the most common problems in pediatrics. Differentiating between bacterial infections, that require antibiotic therapy, and viral infections that resolve on their own is an important challenge for physicians.

C-reactive protein (CRP) is a protein that increases in response to inflammation and its level is generally higher in bacterial infections compared to viral infections. it can be measured by a simple blood test, however its utility as a sole marker for bacterial infection is limited.

The hypothesis of the study is that measuring CRP velocity, e.g the value of CRP divided by the hours since the fever started will improve the utility of CRP for the diagnosis of bacterial infections in children.

ELIGIBILITY:
Inclusion Criteria:

* children less than 5 years of age,
* children with no comorbidities and fever > 38 for at least 24 hours, and
* children with no previous antibiotic therapy.

Exclusion Criteria:

* HIV,
* immunosuppressive conditions,
* antibiotic therapy.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children < 5 years of age presenting to the Emergency Department with fever
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)